CLINICAL TRIAL: NCT02228538
Title: Total Knee Arthroplasty Functional Outcomes Study Research Design
Status: Terminated | Type: Observational
Why Stopped: Not enough subject participation
Sponsor: Restor3D (Industry)
Collaborators: Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 13-003
Record Dates: First submitted 2014-06-05; First posted 2014-08-29 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: total knee arthroplasty; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Arthroplasty, Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total knee arthroplasty patients: ConforMIS iTotal (CR) knee implant system and off-the-shelf knee implant systems from various manufacturers
  Interventions: Device: Total knee arthroplasty patients

INTERVENTIONS:
Device: Total knee arthroplasty patients — ConforMIS iTotal (CR) knee implant system & off-the-shelf standard knee implant system from various manufacturers
  Other Names: knee replacement; joint replacement

SUMMARY:
The purpose of this study is to obtain patient oriented and clinically oriented physical function outcomes both pre-operatively and post-operatively in patients receiving a total knee arthroplasty.

DETAILED DESCRIPTION:
This study aims to use up to 75 patients at 3 centers to determine a baseline short-term post-operative physical function status of patients undergoing a total knee arthroplasty through patient and clinically based assessments. The KOOS score will collect data on the patient's physical function, stiffness and pain. The BERG balance, TUG, and TUDS tests will be used quantitatively to assess the patient's ability to conduct activities of daily living like walking for an extended period of time, standing from a seated position, and maintaining balance while performing a series of actions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or non-pregnant female age 18 years or older at time of study
* Patient is a candidate for a total knee arthroplasty
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation

Exclusion Criteria:

* Patients with a primary diagnosis other than osteoarthritis of the knee as determined by an orthopedic surgeon
* Patients who have had any previous lower extremity procedure
* Patients with a BMI greater than or equal to 40
* Patients with an active infection within the affected knee joint
* Patients with a neuromuscular or neurosensory deficiency that may limit the ability of the patient to evaluate the safety and efficacy of the device
* Patients diagnosed with systemic disease or metabolic disorder leading to progressive bone deterioration (e.g. Lupus Erythematosus, Paget's disease)
* Patients immunologically suppressed or receiving chronic steroids in excess of normal physiological requirements (e.g. greater than 30 days)
* Patients with a known sensitivity to device materials
* Non-English speaking patients
* Patient is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total knee arthroplasty patients
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Timed Functional Tests at 6 weeks | 6 weeks post-op
  Assess patient functional outcomes over time. Comparing times from pre-op to post op of patients performing the same functional tests.
Timed Functional testing at 6 months | 6 months post op
  Assess patient functional outcomes over time. Comparing times from pre-op to post op of patients performing the same functional tests.
Timed Functional Testing at 1 year | 1 year post-op
  Assess patient functional outcomes over time. Comparing times from pre-op to post op of patients performing the same functional tests.

SECONDARY OUTCOMES:
Outcome questionnaires at 6 weeks | 6 weeks post-op
  Assess knee pain and function scores over time. Comparing questionnaire scores from pre-op to post op of patients.
Outcome questionnaires at 6 months | 6 months post-op
  Assess knee pain and function scores over time. Comparing questionnaire scores from pre-op to post op of patients.
Outcome questionnaires at 1 year | 1 year post op
  Assess knee pain and function scores over time. Comparing questionnaire scores from pre-op to post op of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Deryk Jones, MD, Principal Investigator — Ochsner Heath System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States